CLINICAL TRIAL: NCT01112150
Title: Effect of Normatec Pump for Relief of Leg Edema: Short- Intermediate- and Longer-term Outcomes
Brief Title: Effect of Normatec Pump for Relief of Leg Edema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: David S. Blondheim, Hillel Yaffe Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0063-09-HYMC-CTIL
Record Dates: First submitted 2010-04-12; First posted 2010-04-28 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Edema; Heart Failure; Pulmonary Hypertension
Keywords: Edema; Heart failure; Pulmonary hypertension; Edema in legs
MeSH Terms: conditions — Edema; Heart Failure; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pumping group (Active Comparator): Patients in this arm will get a pumping session 2-3 times a day .
  Interventions: Device: NormaTec Pump
- No pumping (Active Comparator): These patients will not receive pumping but only classical treatment clinically indicated (diuretics, oxygen, Digoxin, Nitrates, ACE inhibitors etc, as necessary)
  Interventions: Device: NormaTec Pump

INTERVENTIONS:
Device: NormaTec Pump — Normatec Pump

SUMMARY:
The investigators hypothesize that leg edema will decrease rapidly when using the NormaTec pump, patients will lose weight, will feel better, will be less prone to infections in their legs and to congestion of the liver. Temporary elevation of intravascular fluid volume by the mobilized edema fluid returned to the intravascular space by pumping may increase cardiac output and renal perfusion and in addition it may distend the right atrium and ventricle thus inducing BNP secretion. Both mechanisms may promote excess fluid removal by the kidneys.

ELIGIBILITY:
Inclusion Criteria:

* hemodynamically stable adult patients with pronounced leg edema from any etiology, on optimal medical therapy (such as diuretics, ACE-I or ARBs, digoxin).
* documentation of right heart failure by Echo or other modality (CT, MRI, right heart catheterization) and hemodynamic data from Echo is required and an elevated pulmonary artery pressure (> 35 mmHg) is expected in such cases.

Exclusion Criteria:

* patients in sepsis,
* hemodynamically unstable,
* during an acute attack of pulmonary edema,
* with renal failure (creatinine > 2 mg%),
* with DVT,
* psychiatric or noncompliant patients, and
* patients who will not sign the informed consent form will be excluded from the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 5 days
  The weight loss during the pumping pariod is related to fluid loss from edematous legs.

SECONDARY OUTCOMES:
Leg circumference | 5 Days
  The leg circumference will be measured before and after each pumping session to determine the effectiveness of the pumping.

CONTACTS AND LOCATIONS:
Locations (1):
- Hille Yaffe Medical Ceter, Hadera, Israel, Israel